CLINICAL TRIAL: NCT01750827
Title: A Single Dose Study to Assess the Effect of Non-Bioenhanced, Non-Enteric Coated, Freebase SB-659032 on Platelet Function in Healthy Adult Subjects
Brief Title: A Study to Assess the Effect of SB 659032 on Platelet Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102487
Record Dates: First submitted 2012-12-06; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Atherosclerosis
Keywords: platelet function; atherosclerosis,; SB-659032
MeSH Terms: conditions — Atherosclerosis | interventions — rilapladib

ARMS (1):
- SB-659032 (Experimental): Single dose open label
  Interventions: Drug: SB659032

INTERVENTIONS:
Drug: SB659032 — single dose

SUMMARY:
This will be an open-label, single dose, single period study. Approximately 14 subjects will receive one dose of 250 mg of non-enteric coated SB-659032 following a low-fat breakfast. This study will evaluate whether SB-659032 has an effect on platelet function as determined by platelet aggregation tests using the agonists ADP and collagen. Blood samples for PK analysis and measurement of Lp-PLA2 activity will also be collected

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females who are 18 to 55 years of age, inclusive.
* Body weight greater than 50 kg (110 pounds) and body mass index (BMI) between 19 and 30 where: BMI = weight in kg (height in meters)2

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination or ECG
* History of asthma, anaphylaxis or anaphalactoid reactions, severe allergic responses
* History of smoking within six months of the study and/or has a positive urine cotinine at screening
* History of alcohol consumption exceeding, on average, 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of the first dose of study medication
* Positive urine drug or alcohol at screening
* Use of aspirin, aspirin-containing products, non-steroidal anti-inflammatory agents or any antiplatelet medication within 14 days prior to the first dose of study medication (a list of these drugs will be reviewed with the subject at screening and provided to them to take home)
* Use of prescription (including hormone replacement therapy) or non-prescription drugs and vitamins within 7 days or 5 half-lives (whichever is longer) prior to administration of study medication. An exception is acetaminophen which is allowed at doses of less than and equal to 2g/day for up to 48 hours prior to dosing
* Use of dietary/herbal supplements including (but not limited to) St. John's wort, kava, ephedra (ma huang), gingko biloba, DHEA, yohimbe, saw palmetto, ginseng and red yeast rice within 14 days prior to treatment with study medication
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing
* Consumption of grapefruit or grapefruit juice within 7 days prior to the first dose of study medication
* A history of biliary tract disease including a history of liver disease with elevated liver function tests of known or unknown etiology
* Pregnant or nursing female subjects. For female subjects, a positive serum β-hCG at screening or Day -1; or for female subjects of childbearing potential an unwillingness to agree to one of the methods of contraception listed in the protocol from screening until the completion of follow-up procedures. Hormonal contraceptive methods (e.g. oral contraceptive pill, implant) for female subjects are not permitted. At least a one week interval between screening and first study drug administration will be observed for the pregnancy tests.
* For male subjects, an unwillingness to abstain from sexual intercourse with pregnant or lactating women or an unwillingness to use a condom and another form of contraception (e.g., IUD, birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a woman who could become pregnant until discharge from the study Donation of blood in excess of 500 mL within 56 days prior to dosing
* Full ADP- and/or collagen-induced aggregation (greater than and equal to 40%) at all three concentrations of one or both agonists, as assessed on Day -1
* No ADP- or collagen-induced aggregation (<40%) at the highest concentration of either agonist, as assessed on Day -1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2004-09; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | 24 hours
  Percent maximum platelet aggregation following ADP- and collagen-induced aggregation a 24-hour post-dose period. Other pharmacokinetic endpoints of interest are Tmax of SB-659032 and its pharmacologically active metabolite, SB-664601, as well as Cmax of SB-664601 and concentrations of SB-664601 over a 24-hour post-dose

SECONDARY OUTCOMES:
PK of SB-659032 and SB-664601 | 24 hours
  Cmax of SB-659032 and concentrations of SB-659032 at collection timepoints over
Pharmacodynamics | 24 hours
  Plasma Lp-PLA2 activity, expressed in terms of percent inhibition
Safety/tolerability | 24 hours
  Spontaneous AE reporting, 12-lead ECGs, vital signs, nursing/physician observation, and clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lenexa, Kansas, United States